CLINICAL TRIAL: NCT05210127
Title: Improving the Function of the Foot by Core Foot System (CFS) Exercise Theory in Patients After Hallux Valgus Surgery
Brief Title: Improving the Function of the Foot by Core Foot System (CFS) Exercise Theory in Patients After Hallux Valgus Surgical Procedure
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Józef Piłsudski University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKE 01-42/2021
Record Dates: First submitted 2021-12-01; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2021-11

CONDITIONS: Hallux Valgus
Keywords: hallux valgus; core foot system; rehabilitation protocol
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- After Scarf Osteotomy Group (Experimental): 30 participants after surgery
  Interventions: Procedure: Scarf osteotomy for Hallux Valgus deformity
- Without Scarf Osteotomy Group (Experimental): 30 participants without surgery
  Interventions: Procedure: Scarf osteotomy for Hallux Valgus deformity

INTERVENTIONS:
Procedure: Scarf osteotomy for Hallux Valgus deformity — An experiment of foot muscle strength and activation, during gate phases after hallux valgus correction with the use of core foot system protocol

SUMMARY:
The aim of the study is to identify the impact of CFS foot muscle training on time-space parameters, anthropometric parameters and bioelectrical activity (EMG) of the foot muscles during walking and to develop an algorithm for an effective therapeutic method in patients after hallux valgus correction. Achieving the purpose of the research will contribute to the answer to the following research questions:

* Does the CFS therapy used significantly change the arch of the foot in HV patients compared to the control group?
* Does the CFS therapy used significantly improve gait characteristics after HV surgery in relation to the control group?
* Does muscle stimulation and the moment of their activation differ in groups in which different therapies have been used?
* Will the results of the questionnaires and scale be significantly different in both groups?

ELIGIBILITY:
Inclusion Criteria:

* hallux valgus deformity
* surgical procedure
* voluntary consent to the study

Exclusion Criteria:

* lack of consent to research
* other deformation and operations of the foot
* pain after the surgery which prevents experimental procedure

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
American Orthopaedic Foot and Ankle Scale for first metatarsophalangeal joint | 8 weeks
  Orthopaedic Scale to describe function and problems with first metatarsophalangeal joint
The 36-Item Short Form Survey (SF-36) | 8 weeks
  The SF-36 is often used as a measure of a person or population's quality of life (QOL)
Zebris Medical System | 8 weeks
  The plantar pressure distribution measurement systems
EMG test | 8 weeks
  Electromyography (EMG) measures muscle response or electrical activity in response to a nerve's stimulation of the muscle
Podoscope test | 8 weeks
  A diagnostic device that allows the assessment of the sole of the foot while standing

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Baran M, Kolodziejski P, Kaczmarczyk K. Protocol: a randomized parallel-group study of women after hallux valgus correction surgery to compare the effects of "core foot system" training vs. traditional rehabilitation methods. Acta Bioeng Biomech. 2024 Feb 26;25(4):103-109. doi: 10.37190/abb-02332-2023-03. Print 2023 Dec 1. PMID 39072466